CLINICAL TRIAL: NCT03732378
Title: Role of Omega-3 Polyunsaturated Fatty Acid in the Management of Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allama Iqbal Open University Islamabad (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Naiza Yousef, Nutritionist, Allama Iqbal Open University Islamabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 561/17
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Role of Omega-3 Polyunsaturated Fatty Acid in the Management of Major Depressive Disorder: A Randomized Controlled Trial
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: 12 week Randomized, single blind, placebo-Controlled Trial (RCT) was conducted at King Edward medical university, psychiatry & behavioral sciences department Lahore. one capsule of omega-3 (EPA 300mg, and 200mg DHA) were given, or placebo (500 mg corn oil).
Who Masked: Participant
Masking Description: Along with anti psychotics, one capsule of omega-3 (EPA 300mg, and 200mg DHA) were given to treatment group , and 500 mg corn oil one capsules daily along with anti psychotics were given to placebo group. Patients were unaware about treatment and placebo as plastic transparent same packing was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-3 (Experimental): one capsule of omega-3 (EPA 300mg, and 200mg DHA) were given to treatment group along with already taking anti depressant drugs( citalopram, escitalopram, paroxetine 1 tablet at night time)
  Interventions: Dietary Supplement: Omega-3 capsule
- Placebo (Placebo Comparator): one capsule of 500 mg corn oil, along with already taking anti depressant drugs( citalopram, escitalopram, paroxetine 1 tablet at night time) were given to placebo group
  Interventions: Dietary Supplement: Omega-3 capsule

INTERVENTIONS:
Dietary Supplement: Omega-3 capsule — Daily one capsule of omega-3 (EPA 300mg, and 200mg DHA) were given anti depressent( citalopram, escitalopram, paroxetine 1 tablet at night time)

SUMMARY:
Background: Patients with major depressive disorder have prominently been reported to be related with subnormal polyunsaturated omega-3 fatty acids levels, importantly low docosahexaenoic acid and eicosapentaenoic acid in plasma and dietary intake. However, more randomized controlled trials are needed to support its importance in management of depression.

Objective: To explore polyunsaturated omega-3 fatty acid role in major depressive disorder management.

Materials & Methods: Seventy patients 20 to 40 yeas, who were already diagnosed with depression and taking antidepressant treatment, were selected at department of psychiatry and behavioral sciences Kind Edward Medical University Lahore, and assigned into 2 groups, i.e. Intervention and control, by simple random lottery method. For twelve weeks, intervention group advised to take one omega-3 (300mg EPA, eicosapentaenoic acid and 200mg DHA docosahexaenoic acid), or placebo (500 mg corn oil) capsules once daily with meal. Beck Depression Inventory (BDI) scale was used to assess the depression. Demographic information was collected by using a structured questionnaire.

DETAILED DESCRIPTION:
Study Design:

12 week Randomized, single blind, placebo-Controlled Trial (RCT) was conducted at King Edward medical university, psychiatry & behavioral sciences department Lahore. From 19 May 2017 to 16 August 2017 one capsule of omega-3 (EPA 300mg, and 200mg DHA) were given (38, 39), or placebo (500 mg corn oil) (40).

Data Collection and Evaluation:

Subjects were assessed at the first visit according to inclusion and exclusion criteria. Information about demographics, dietary habits and risk factors such as age, gender, height, weight and family history of depression, dietary habits, education levels, marital status, cigarette smoking, supplementation and sleeping hours were obtained by using a structured questionnaire in face to face interview in local and easy to understand language. BMI was calculated by using the equation BMI=kg/m2.

Ethical Approval:

Written approval (Reg.No.Psy/561/17) was taken from the head of psychiatry & behavioral sciences department, King Edward medical university Lahore. Informed consent had been taken from all study participants in written form after explaining the procedure of the study. Guidelines laid out in the Declaration of Helsinki were followed to conduct this study.

Statistical Analysis:

Data was analyzed through SPSS 20.0 with 95% confidence interval. Frequency distribution and of demographic variables were checked. Chi square test was used to check the relationship between depression and risk factors. Paired T test was used to analyze the before and after intervention mean difference. Results were presented in tabular and graphical form.

ELIGIBILITY:
Inclusion Criteria:

Patient aged from 20 to 40 years age and taking anti-depressant drugs, were selected for study.

Exclusion Criteria:

Pregnant and lactating women and patients with history of allergy to omega-3 fatty acids shellfish were excluded.

Patients with Serious neurological and medical conditions that can likely to interfere with the treatment of depression such as dementia, schizophrenia, epilepsy were also excluded.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Beck depression inventory scale | half an hour
  Normal ups down (1-10) Mild mood disturbance (11-16) Borderline clinical depression (17-20) Moderate depression (21-30) Severe depression (31-40) Extreme depression (over 40)

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Ahmad, Phd, Study Director — Allama Iqbal Open University Islamabad
Locations (1):
- Zaheer Ahmad, Islamabad, Punjab Province, Pakistan

REFERENCES:
- [Background] Arnaud A, Gayrard P, Ohresser P. [Bronchomotor tonus: per-operative bronchospasm]. Ann Anesthesiol Fr. 1976;17(2):139-44. French. PMID 62529
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851